CLINICAL TRIAL: NCT06462573
Title: Extra-Corporeal Shock Wave Lithotripsy for Renal and Upper Ureteral Stones in Adults Under Locally Infiltrate d Anaesthetics ; a Clinical Randomized Controlled Study
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hosam salah abd elrahim, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Eswl
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Stone Ureter
MeSH Terms: conditions — Ureterolithiasis | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (study group) (Experimental): in which patients will undergo ESWL under locally infiltrated anaesthetic. Using ultrasound guidance, the quadratus lumborum muscle will be identified. Then a mixture of 0.5 % bupivacaine (10 ml) and 2 % lidocaine (10 ml) will be injected into the muscle as a single shot 20 minutes before the procedure.
  Interventions: Drug: locally infilterating anaethesia like lidocaine
- Group II (control group) (Experimental): in which patients will undergo ESWL under systemic analgesia. The latter will be achieved using one gram of paracetamol IV infusion at the beginning of the procedure.
  In case of unsatisfactory pain control in either group, systemic analgesia using IV Ketorolac injection will be used on demand or the required dose will be recorded at the end of the session.
  Interventions: Drug: general anaethesia

INTERVENTIONS:
Drug: locally infilterating anaethesia like lidocaine — which patients will undergo ESWL under locally infiltrated anaesthetic. Using ultrasound guidance, the quadratus lumborum muscle will be identified. Then a mixture of 0.5 % bupivacaine (10 ml) and 2 % lidocaine (10 ml) will be injected into the muscle as a single shot 20 minutes before the procedure.
  Other Names: Group I (study group)
  Arms: Group I (study group)
Drug: general anaethesia — which patients will undergo ESWL under systemic analgesia. The latter will be achieved using one gram of paracetamol IV infusion at the beginning of the procedure.
  In case of unsatisfactory pain control in either group, systemic analgesia using IV Ketorolac injection will be used on demand or the required dose will be recorded at the end of the session.
  Other Names: Group II (control group)
  Arms: Group II (control group)

SUMMARY:
There are many treatment modalities available for managing renal and upper ureteric stones. They range from completely non-invasive outpatient procedures to invasive procedures requiring hospital admission and increased risks of complications. Extracorporeal shockwave lithotripsy (ESWL) is a truly non-invasive procedure as opposed to other surgical treatments used, such as retrograde intrarenal surgery and percutaneous nephrolithotomy (1).

The choice between shockwave lithotripsy (SWL) and other treatment modalities depends on several factors, including stone site, stone burden, stone CT density, etc. Another compounding factor in choosing the treatment modality is patient preference and expectation (1).

Extracorporeal Shock Wave Lithotripsy is one of the treatment options for patients with renal and ureteral calculi. Even though the procedure is less invasive compared to others. Pain caused by the procedure is a major concern. Several studies recommended the use of either local or systemic analgesia with varying results (2).

As a truly non-invasive treatment option, ESWL has been widely used for treating renal, as well as ureteric, stones with satisfactory efficacy and minimal morbidity. However, the pain caused by ESWL is a major limitation of its efficacy, in addition to the associated patient dissatisfaction and negative experience that may result in the patient refraining from further sessions.

The relationship between pain and ESWL efficacy can be explained by multiple facts: firstly, the pain leads to inability to increase the energy delivered by the shockwaves to optimum levels; secondly, the pain usually leads to significant movement of the patient, as well as excessive respiratory movements, both of which move the stone away from the focus of shockwaves; lastly, the pain may be severe that the session is discontinued before delivery of effective number of shockwaves

DETAILED DESCRIPTION:
There are many treatment modalities available for managing renal and upper ureteric stones. They range from completely non-invasive outpatient procedures to invasive procedures requiring hospital admission and increased risks of complications. Extracorporeal shockwave lithotripsy (ESWL) is a truly non-invasive procedure as opposed to other surgical treatments used, such as retrograde intrarenal surgery and percutaneous nephrolithotomy (1).

The choice between shockwave lithotripsy (SWL) and other treatment modalities depends on several factors, including stone site, stone burden, stone CT density, etc. Another compounding factor in choosing the treatment modality is patient preference and expectation (1).

Extracorporeal Shock Wave Lithotripsy is one of the treatment options for patients with renal and ureteral calculi. Even though the procedure is less invasive compared to others. Pain caused by the procedure is a major concern. Several studies recommended the use of either local or systemic analgesia with varying results (2).

As a truly non-invasive treatment option, ESWL has been widely used for treating renal, as well as ureteric, stones with satisfactory efficacy and minimal morbidity. However, the pain caused by ESWL is a major limitation of its efficacy, in addition to the associated patient dissatisfaction and negative experience that may result in the patient refraining from further sessions.

The relationship between pain and ESWL efficacy can be explained by multiple facts: firstly, the pain leads to inability to increase the energy delivered by the shockwaves to optimum levels; secondly, the pain usually leads to significant movement of the patient, as well as excessive respiratory movements, both of which move the stone away from the focus of shockwaves; lastly, the pain may be severe that the session is discontinued before delivery of effective number of shockwaves

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older whether males or females with renal or upper ureteric stone(s) candidate for ESWL therapy 2. Renal stones should be between 1- 2 cm and upper ureteric stones should be less than 15 mm

Exclusion Criteria:

* 1.. Patients refusing to participate in the study or patients not compliant with follow up 2. Renal stones in ectopic kidneys 3. Radiolucent upper ureteric stones 4. Patients with myo-skeletal deformities e.g. kyphoscoliosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between local and systemic analgesia | Baseline
  Pain score during the session using visual analogue scale

SECONDARY OUTCOMES:
Comparison between local and systemic analgesia | Baseline
  4. Two-month stone free rate (SFR)

CONTACTS AND LOCATIONS:
Overall Officials: Salah El-Din Shaker Abdel Hafez, Study Director — professor; Nasreldin Abdelaal, Study Director — assistant professor

REFERENCES:
- [Background] Manzoor H, Leslie SW, Saikali SW. Extracorporeal Shockwave Lithotripsy. 2024 Oct 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK560887/ PMID 32809722
- [Background] Laksita TB, Soebadi MA, Wirjopranoto S, Hidayatullah F, Kloping YP, Rizaldi F. Local anesthetics versus systemic analgesics for reducing pain during Extracorporeal Shock Wave Lithotripsy (ESWL): A systematic review and meta-analysis. Turk J Urol. 2021 Jul;47(4):270-278. doi: 10.5152/tju.2021.21143. PMID 35118950
- See also: personal email — http://hossalah111@gmail.com